CLINICAL TRIAL: NCT04953806
Title: The Development of an Integrated Physical Activity and Mental Health Intervention for Veterans With COPD, Emotion Distress, and Low Physical Activity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3527-W
Record Dates: First submitted 2021-06-24; First posted 2021-07-08 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: COPD; Depression; Anxiety
Keywords: COPD; Physical Activity; Depression; Anxiety
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Depression; Anxiety Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: Assess the feasibility of Step-CBT in a proof-of -concept, single-arm trial in Veterans (Enrollment target; N=40) with COPD, low physical activity, and clinically significant depression and/or anxiety symptoms. Targeting 25 completers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Step-CBT (Experimental): Participants will complete Step-CBT, an integrative 8-week physical activity and cognitive behavioral therapy (CBT) intervention, delivered by a licensed clinical psychologist. Sessions will take place once per week for 60 minutes using VA Video Connect. Each session will include core components 1) Reviewing physical activity goals, prescribing new step count goal, and problem-solving barriers and 2) The weekly CBT intervention module.
  Interventions: Behavioral: Step-CBT

INTERVENTIONS:
Behavioral: Step-CBT — Participants will complete Step-CBT, an integrative 8-week physical activity and cognitive behavioral therapy (CBT) intervention, delivered by a licensed clinical psychologist. Sessions will take place once per week for 60 minutes using VA Video Connect. Each session will include core components 1) Reviewing physical activity goals, prescribing new step count goal, and problem-solving barriers and 2) The weekly CBT intervention module.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is prevalent and debilitating chronic disease in Veterans. COPD is highly co-morbid with depression and anxiety conferring greater morbidity and mortality risk. Physical activity is a modifiable behavior that can improve COPD outcomes. However, to date, interventions targeting physical activity have not addressed the high comorbidity between COPD and depression and/or anxiety symptoms ("emotional distress") despite emotional distress predicting poorer response to physical activity interventions. This CDA-2 proposal will develop and test the acceptability and feasibility of an integrative physical activity and mental health intervention for Veterans with COPD, emotional distress, and low physical activity. The intervention will be delivered via VA Video Connect enabling access to care among Veterans with substantial barriers to hospital-based outpatient care.

DETAILED DESCRIPTION:
The current study will develop and test Step-Cognitive Behavioral Therapy (CBT) (Step-CBT), an integrated intervention that draws from existing pedometer-based physical activity (PA) interventions and brief CBT to target low PA, emotional distress, and physical disability in Veterans with chronic obstructive pulmonary disease (COPD) delivered via VA Video Connection (VVC). This study has three components: In Aim 1, we will conduct a cross-sectional study with 50 Veterans with COPD, low PA, and clinically significant depression and/or anxiety symptoms. Self-report measures will be collected and provide information on mean level and magnitude of the relations between PA, emotional distress, and physical disability. Participants will wear an ActiGraphy device for 14 days following their in-person session to measure objective PA. Based on these data, we will create Step-CBT, an intervention that integrates, tailors, and adapts a pedometer-based PA intervention and brief CBT (existing transdiagnostic protocol), based on patient interviews and current literature. In Aim 2, we will examine the acceptability of Step-CBT, an 8-session intervention delivered via VVC, in Veterans (N=6) collecting recruitment, enrollment, completion data and measures of physical functioning and emotional distress. We will conduct expert panel review of the manualized intervention protocol and acceptability results. In Aim 3, we will assess the feasibility of Step-CBT in a proof-of -concept study design in Veterans (N=40 enrolled with target of 25 completers) with COPD, low physical activity, and clinically significant depression and/or anxiety symptoms. The current research has great potential to improve physical and psychological functioning in Veterans with COPD through the development of an integrated PA-mental health intervention. Step-CBT delivered to patient's homes, would offer a safe option to increase/maintain physical functioning and mental health in Veterans with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Any gender-identified, greater than or equal to 40 years of age
* Clinical diagnosis of COPD defined as the presence of emphysema on a CT scan and one piece of clinical evidence of COPD (defined as a ratio of FEV1 to forced vital capacity < 0.70, > 10 pack-year cigarette smoking history, overall assessment of COPD in their problem list or in Pulmonary/Primary Care notes, or on bronchodilators (specifically antimuscarinics such as Tiotropium or Ipratropium). If there is no evidence of emphysema, or no CT on scan in their medical chart, three pieces of clinical evidence of COPD will suffice for a clinical diagnosis of COPD.
* Ability to communicate
* Able to participate in in-person study appointment at the VA
* English speaking
* Competent to provide informed consent
* Emotional distress. Clinically significant depression and/or anxiety defined as PHQ-8 > 10 and/or Beck Anxiety Inventory > 13
* Wireless Internet connection and Bluetooth capability
* Participants with > 90% accuracy of device Fitbit to manual step counts
* Agreeable to audio record study session
* Agreeable to wearing an ActiGraphy device and Fitbit and downloading the Fitbit app
* Email user for VVC visits links
* Either owns a smartphone or iPad compatible with the Fitbit app and enabled with Bluetooth or agreeable to using a study-issued iPad with Wi-Fi and Bluetooth capabilities
* Medical clearance from healthcare provider to participate in a physical activity program

Exclusion Criteria:

* COPD exacerbation in the previous 1 month
* Inability to ambulate
* Regular use of a rollator, walker, or wheelchair for ambulation
* Inability to complete questionnaires
* Inability to collect at least 4 valid days of 7-day baseline step count data
* Positive screening on the Mini-Cog defined as < 3 indicating possible cognitive impairment or dementia or major neurocognitive disorder diagnosis in electronic medical chart or refusal to complete the assessment
* Currently enrolled in another interventional study targeting exercise, physical activity, or mental health
* Average baseline step counts of greater than or equal to 10,000 steps per week
* Suicide flag in chart
* Oxygen saturation after 6-Minute Walk Test documented to be <85%

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Measuring change - Late Life Function and Disability Instrument (LLFDI) | Baseline, Week 8 (mid-point), Week 16 (post-intervention) - measuring change
  Change in scores on the Late Life Function and Disability Instrument (LLFDI) from baseline to Week 15. The LLFDI is a 32-item measure of self-reported functional impairment and disability. Respondents indicate the degree of difficulty they have performing physical activities without the help of someone or using assistive devices. Scores range from 0 to 100 with higher scores indicating higher levels of functioning. We will only use the Disability component of the LLDFI. The LLDFI is sensitive to change and commonly used as an outcome in geriatric research.
Step Count-measuring change | Baseline, Week 8 (mid-point), Week 16 (post-intervention)- measuring change
  Change in Step Count. We reference prior MID for estimates of change: Minimally Important Difference = 600-1000 steps. Step count will be measured using two devices:
  The ActiGraph wGT3X-BT. The ActiGraph wGT3X-BT is research-grade, highly accurate measure of activity, through the use of a special sensor detecting acceleration, position, and timing, to detect steps. The device is worn around the ankle and is unobtrusive.
  - The FitBit Inspire serves as a tool to track and monitor step counts weekly as part of the intervention and to develop weekly step count goals.
  Both methods of measuring step count will be reported.

SECONDARY OUTCOMES:
Patient Health Questionniare-8- measuring change | Baseline, Week 8 (mid-point), Week 16 (post-intervention)- measuring change
  Change in scores on the Patient Health Questionnaire-8 (PHQ-8) from baseline to Week 16. The PHQ-8 is an 8-item measure of depression symptoms severity mapping on to DSM-IV criteria. Higher scores are indicative of more severe depression symptoms. Score range from 0 to 24, with higher scores indicative of greater depression symptom severity. We use estimates of clinically meaningful change in the literature: PHQ-8 (≤9 combined with improvement of 50%).
  Meaningful change in the literature is PHQ-9 score (< = 9 combined with improvement of 50%). The PHQ-9 is a 9-item measure of depression symptoms severity mapping on to DSM-IV criteria. Higher scores are indicative of more severe depression symptoms. Score range from 0 to 27, with higher scores indicative of greater depression symptom severity.
Beck Anxiety Inventory- measuring change | Baseline, Week 8 (mid-point), Week 16 (post-intervention)- measuring change
  Change in scores on the Beck Anxiety Inventory (BAI) from baseline to Week 16. Meaningful change in the literature is a 17.5% reduction in BAI scores over time. The BAI is a 21-item screening measure of cognitive and somatic symptoms of anxiety over the past week. Respondents indicate the degree to which they experienced each symptom from 0 (not at all) to 3 (severely), ranging from 0 to 63. Higher scores indicated greater anxiety severity.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Bamonti, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No